CLINICAL TRIAL: NCT06557707
Title: Cardiovascular Health & Early Stress
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20021768
Record Dates: First submitted 2024-05-30; First posted 2024-08-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood is collected for routinary biomarkers and exploratory biomarkers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Young individuals ACE (ages 18-30 years old): Young individuals who experienced accumulative adverse childhood experiences
  Interventions: Other: Childhood stress
- Children ACE (ages 9-17 years old): Children who experienced accumulative adverse childhood experiences .
  Interventions: Other: Childhood stress
- Young individuals No ACE (ages 18-30 years old): Young individuals who have not experienced accumulative adverse childhood experiences
- Children No ACE (ages 9-17 years old): Children who have not experienced accumulative adverse childhood experiences.

INTERVENTIONS:
Other: Childhood stress — Based on stress-related information, participants will be divided into those who were exposed to adversity during childhood and those who were not exposed.
  Groups: Children ACE (ages 9-17 years old); Young individuals ACE (ages 18-30 years old)

SUMMARY:
Childhood adversity is highly prevalent, with 59% of the U.S. population reporting at least one adverse childhood experience (ACE). Substantial evidence links childhood adversity to cardiometabolic disease later in the life course, including heart disease, diabetes, and stroke, which are 3 of the top 10 causes of mortality in the United States.

ACEs encompass many possible traumatic and distressing experiences, including abuse, neglect, or severe household dysfunctions. It is not surprising that the experience of those extreme events during the first decade of life has tremendous implications for the individual's psychological and physical health.

DETAILED DESCRIPTION:
Current knowledge supports that ACEs trigger emotional stress, anxiety, fear, and discomfort in the individual. Acute and intense mental stress leads to structural changes in the amygdala, prolonged activation of the hypothalamic-pituitary-adrenal axis, and hyperactivation of the sympathetic nervous system. Then, the body secretes hormones to activate the cardiovascular system to cope with stress with a rapid increase in arterial pressure and heart rate. If the trauma is severe and/or repeated, the resting state for heart rate and blood pressure are readjusted, resulting in these children living in a heightened physiological state of arousal, including higher heart and respiration rates. This status leads to endothelial dysfunction and atherothrombotic activation that can contribute to premature cardiovascular dysfunctions. Notably, there is evidence of a cumulative effect, or dose-response relationship, between the number of reported ACEs and the prevalence of health risk behaviors and chronic diseases. Thus, despite the prevalence of ACEs and the impact on health and society, the mechanisms underlying these dysfunctions are still poorly understood. The present study aims to understand the impact of different types of ACEs on cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* Men and pre-menopausal women
* 18-30 years old

Cohort 2

* males and females
* 9-17 years old

Exclusion Criteria:

Cohort 1

* Evidence of cardiovascular, pulmonary, renal, hepatic or cerebral diseases
* Evidence of pregnancy or currently nursing.
* Having a history of chronic pain
* Having a history of rheumatoid arthritis

Cohort 2

* Evidence of cardiovascular, pulmonary, renal, hepatic or cerebral diseases
* Evidence of pregnancy or currently nursing.
* Having a history of chronic pain
* Having a history of rheumatoid arthritis

Ages: 9 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and young individuals who have been exposed to adversity during childhood
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Vascular function | Baseline
  This test examines how the blood vessels respond to different challenges and expand. It is used to characterize the cardiovascular health of the subject's blood vessels. Different events and substances will be used (under an IND) to test how the blood vessels react. The test is completed using Laser Doppler Speckle Contrast. We will measure how much the blood vessels dilate. Greater dilation, better vascular function.
Cardiac Function | Baseline
  An evaluation of cardiac response will be monitored non-invasively. We will use ultrasound to visualize the heart and the blood vessels.
Cardiac MRI (CMR) | Baseline
  Cardiac MRI will be completed to monitor early signs of poor functionality.

SECONDARY OUTCOMES:
Spirometry | Baseline
  Subjects will undergo a lung function test to measure how well their lungs work. The volume of air moving in and out of the lungs will be assessed. FEV1 will be evaluated. FEV1 is the amount of air a person can exhale in the first second after inhaling as deeply as possible.
Lung Diffusing Capacity | Baseline
  Subjects will undergo a lung function test to measure how well their air is diffused from their lungs. DLCO will be evaluated. DLCO stands for diffusing capacity of the lungs for carbon monoxide, and it's a pulmonary function test that measures how well oxygen moves from the lungs into the bloodstream.
Complete blood count | Baseline
  Blood analysis
HbA1c | Baseline
  Blood analysis
C-Reactive protein | Baseline
  Blood analysis
Questionnaires | Baseline
  Lifestyle and stress related questionnaires will be completed by the participants including lifestyle, adversity during childhood, stress risk.
Arterial Stiffness | Baseline
  A non-invasive assessment will be used to measure how fast the participant's blood travels, which is a measure of how stiff their arteries are.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rodriguez Miguelez, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States